CLINICAL TRIAL: NCT07040007
Title: The Effects Of Balance Exercises Versus Strengthening Exercises On Gait And Cognitive Parameters In Geriatric Individuals With Early-Stage Dementia
Brief Title: Comparison of Strengthening and Balance Exercises in Early-Stage Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Beyza Kuşva (Other)
Responsible Party: Sponsor-Investigator, Zeynep Beyza Kuşva, Master's Student Researcher, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/259
Record Dates: First submitted 2025-06-11; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Physical Therapy
Keywords: dementia; exercise; gait; cognitive function
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Exercise (Experimental)
  Interventions: Behavioral: Balance Exercises
- Strengthening Exercise (Experimental)
  Interventions: Behavioral: Strengthening Exercises

INTERVENTIONS:
Behavioral: Strengthening Exercises — In the strengthening exercises, the amount of weight was determined based on 40 to 60 percent of the one-repetition maximum. Each exercise was performed in two sets of six to eight repetitions. The exercise sessions lasted approximately 40 minutes and included a 10-minute warm-up, 20 minutes of strengthening exercises, and a 10-minute cool-down period. To perform the strengthening exercises, resistance bands (Theraband), dumbbells, weighted balls, sandbags, and a resistance bicycle were used. The exercises were performed for both the upper and lower extremities.
  For the upper extremities, shoulder abduction, elbow extension, and shoulder extension exercises were performed using a theraband; elbow flexion, shoulder flexion, and elbow extension exercises were performed using dumbbells; and shoulder abduction exercises were performed using a weighted ball. For the lower extremities, knee extension, hip extension, and hip abduction exercises were performed using a resistance bicycle.
  Other Names: Group I
  Arms: Strengthening Exercise
Behavioral: Balance Exercises — Each session was carried out over approximately 40 minutes, consisting of a 10-minute warm-up, 20 minutes of balance exercises, and a 10-minute cool-down period. The exercises were individually planned based on the participant's performance. To perform the balance exercises, supportive equipment such as balance discs and Pilates balls, as well as environments such as soft surfaces and stairs, were used.
  The balance exercises applied during the intervention included standing on a balance disc with weight shifting, walking on a soft surface, tandem walking, walking while stepping over obstacles, and cross-step walking. Additionally, seated balance activities, standing trunk rotations using a Pilates ball, sit-to-stand exercises from a chair, and stair climbing exercises were also performed as part of the program.
  Other Names: Group II
  Arms: Balance Exercise

SUMMARY:
The aim of this study was to examine and compare the effects of balance exercises versus strengthening exercises on gait and cognitive parameters in older adults with early-stage dementia.

A total of 35 older adults with early-stage dementia were included in the study, and it was completed with 32 participants. The participants were divided into two groups and followed for 8 weeks. Group I received strengthening exercises, while Group II received balance exercises. After recording the demographic and clinical characteristics of all participants, gait was evaluated using the Berg Balance Scale (BBS), spatiotemporal gait parameters, and the Timed Up and Go (TUG) test; cognitive parameters were assessed with the Montreal Cognitive Assessment (MoCA) and the Dynamic Lowenstein Occupational Therapy Cognitive Assessment - Geriatric Version (DLOTCA-G); muscle strength was measured using Activforce-2; and quality of life was evaluated using the WHOQOL-OLD (World Health Organization Quality of Life - Older Adults Module).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65 and 95 years,
* Able to walk 10 meters independently,
* Scoring between 16 and 26 on the Mini Mental State Examination,
* Literate individuals (able to read and write).

Exclusion Criteria:

* Having uncontrolled heart disease,
* Body mass index (BMI) below 18.5 kg/m² or above 35 kg/m²,
* Diagnosed with cancer,
* Completely lost vision,
* Having any disease that may prevent performing exercise.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Balance Performance Assessed by the Berg Balance Scale After 8 Weeks of Treatment | 8 Weeks
  It is scored from 0 to 56, with higher scores indicating better balance performance.
Change from Baseline in Gait Parameters Assessed by Temporal-Spatial Variables After 8 Weeks of Treatment | 8 Weeks
  Within the scope of the Temporal-Spatial Variables Method, step length, double step length, step width, and the number of steps taken per minute were evaluated. Increases in step length and double step length, a decrease in step width, and an increase in the number of steps per minute were associated with improvements in gait.
Change from Baseline in Gait Performance Assessed by the Timed Up and Go Test After 8 Weeks of Treatment | 8 Weeks
  The Timed Up and Go Test is performed by measuring, in seconds, the time it takes for an individual to stand up from a chair, walk 3 meters, turn around, walk back, and sit down again. A shorter time indicates better gait performance.
Change from Baseline in Cognitive Function as Measured by the Montreal Cognitive Assessment (MoCA) After 8 Weeks of Treatment | 8 Weeks
  Cognitive function in the Montreal Cognitive Assessment (MoCA) is scored between 0 and 30, with higher scores indicating better cognitive performance.
Change from Baseline in Cognitive Function as Measured by the Dynamic Loewenstein Occupational Therapy Cognitive Assessment - Geriatric Version (DLOTCA-G) After 8 Weeks of Treatment | 8 Weeks
  The Dynamic Loewenstein Occupational Therapy Cognitive Assessment - Geriatric Version (DLOTCA-G) is a cognitive assessment tool scored between 17 and 119. Higher scores indicate better cognitive functioning.

SECONDARY OUTCOMES:
Change from Baseline in Muscle Strength as Measured by the Activforce 2 Dynamometer After 8 Weeks of Treatment | 8 Weeks
  Activforce-2 is a digital dynamometer used for the objective measurement of muscle strength. In this study, muscle strength of the Biceps, Triceps, Middle Deltoid, Quadriceps, Hamstrings, Gluteal muscles, and Gastrocnemius was assessed using the Activforce-2 device.
Change from Baseline in Quality of Life as Measured by the World Health Organization Quality of Life - Older Adults Module (WHOQOL-OLD) Questionnaire After 8 Weeks of Treatment | 8 Weeks
  The World Health Organization Quality of Life - Older Adults Module (WHOQOL-OLD) is an assessment scale scored between 24 and 120. However, since higher scores in certain items may reflect lower quality of life, it is important to evaluate the individual item scores rather than relying solely on the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep B Kuşva, Principal Investigator — Istanbul University - Cerrahpasa; Ela TARAKCI, Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided